CLINICAL TRIAL: NCT03233503
Title: Taste, Fat Sensation and Texture Study of Dutch and Malaysian Diets
Brief Title: Taste, Fat Sensation and Texture Study
Status: Completed | Type: Observational
Sponsor: Wageningen University (Other)
Collaborators: Taylor's University (Other)
Responsible Party: Principal Investigator, Monica Mars, Dr., Wageningen University
Other Study IDs: NL47315.081.13
Record Dates: First submitted 2017-07-20; First posted 2017-07-28 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Taste Perception; Fat Sensation; Eating Rate; Bite Size

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (2):
- Dutch trained taste panel: The study population consists of a sample of 15 healthy Dutch males and females, recruited in the Wageningen area.
  Interventions: Diagnostic Test: Basic taste, fat sensation and texture perception
- Malaysian trained taste panel: The study population consists of a sample of 20 healthy Malaysian males and females, recruited in the Subang Jaya, Selangor area.
  Interventions: Diagnostic Test: Basic taste, fat sensation and texture perception

INTERVENTIONS:
Diagnostic Test: Basic taste, fat sensation and texture perception — This is an observational Sensory study methodologically similar to "Astringency and bitterness perception clinicalTrials.gov identifier NCT03171402 "Participants are first involved in sensory training sessions that train how they recognise between different basic tastes and differentiate perceived intensity in solutions and foods. After 6 months of training, the trained participants are involved in tasting a wide array of commonly consumed foods. At this study phase, participants will rate for the foods' taste, fat sensation perception and texture

SUMMARY:
Food is selected primarily on their taste and texture properties. It is essential to get more insight in taste and texture characteristics of the foods in the Dutch and Malaysian diets for a better understanding of food choices. Currently, there is insufficient information on taste and texture properties of foods to relate these properties to the composition of diets and individual food choice in larger (observational) studies.

In the current study, the investigators want to assess the perceived intensities of the 5 basic tastes, i.e. sweet, salt, sour, bitter and umami, as well as fat sensation and texture, in an array of about 1,000 often consumed Dutch and Malaysian foods. The investigators aim to do this with a trained sensory panel, which is a well-accepted way of assessing perception of sensory attributes.

With the current study, the investigators aim to build a table, which is comparable to the food composition table, but contains data that describes foods and meals in terms of sensory properties. That is, investigators want to quantify sensory characteristics of about 1,000 commonly eaten Dutch and Malaysian foods. This enables investigators to add sensory information to the food intake data that is already being collected in observational studies, and to further understand food choices in specific populations, such as elderly and patient groups. In current project, the investigators also aim to compare the Dutch diet to the Malaysian diet in term of sensory properties.

DETAILED DESCRIPTION:
The study is an observational study on taste and texture of commonly consumed Dutch and Malaysian foods with three phases, i.e. screening, training and tasting sessions.

The study will be held in the sensory tasting rooms at Wageningen University, The Netherlands and Taylor's University, Malaysia, respectively.

After the recruitment and prior to the training and tasting sessions, there will be a 2-hour screening session (Phase I) during which the investigators will select respective Dutch and Malaysian participants based on their performance in a sensory test.

During the training session (Phase II), the participants need to commit and involve in 2 1½-hour sessions a week for approximately four- six months (until sufficiently trained).

At the tasting sessions (Phase III), trained Dutch and Malaysian panellist also need to involve in 2-3 sessions a week for a consecutive three years. Each session will take approximately 1½ hour. During this session, series of food will be rated for their taste, fat and texture. In addition, food texture will be measured by eating rate and quantifying the size of the bites which it is eaten.

The usual performance of the panellist also are discussed with the panellists and monitored throughout the training phase and regularly (each month) during the tasting phase.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-55 years
* BMI: 18.5-25kg/m2 (self-reported)
* Physically and mentally healthy as not suffering or under control by any medications
* Available during the whole period and shown to be committed to participate 3 times/wk
* Good performance on the sensory tests during the screening

Exclusion Criteria:

* Smoking (equal or more than 1 unit per day and those stopped smoking less than3 months)
* Excessive alcoholic consumer (more than 21 units per week)
* Being vegetarian or having religious dietary restrictions
* Reported to have certain dental limitations (denture, tongue piercing or difficulties in chewing and swallowing)
* Reported intolerance or allergies to foods
* Using medications that are known to affect taste and smell identification
* Being pregnant or lactating
* Participating and/or planning to participate in other studies for the coming three years

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Only Dutchs are allowed to participate as Dutch taste panel; and only Malaysians are allowed to participate as Malaysian taste panel
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2014-03-13 (Actual); Primary Completion 2016-12-22 (Actual); Study Completion 2016-12-22 (Actual)

PRIMARY OUTCOMES:
Comparison of panel performance results of two trained Dutch and Malaysian panelist | Phase II training , an average of 3 hours visit per week
  For individual taste attributes of the reference solutions and reference foods, analysis of variance (ANOVA) was used to evaluate the performance of each panel on discrimination, repeatability and agreement according to the following model:
  Attribute= µ + product (P) + assessor (A) + replicate (r) + product*assessor (P*A) + product*replicate (P*r) + assessor*replicate (A*r) + E, where product= discrimination, assessor= consistency of ratings between assessors, replicate= consistency of ratings from one session to another, product*replicate= panel repeatability, product*assessor = agreement between assessors, assessor*replicate= assessor repeatability. The replicate scores deviated from the product mean for all taste attributes from the total scale were also reported as root mean squared error (RMSE) of the ANOVA model without replicate effect
Dutch trained panelist-generated taste intensity ratings of commonly consumed Dutch foods | Through study completion, an average of 3hours visit per week
  The intensity rating of taste: sweet, salt, sour, bitter, umami and fat sensation on the 100-point quantitative Spectrum scales
Malaysian trained panelist-generated taste intensity ratings of commonly consumed Malaysian foods | Through study completion, an average of 3hours visit per week
  The intensity rating of taste: sweet, salt, sour, bitter, umami and fat sensation on the 100-point quantitative Spectrum scales

SECONDARY OUTCOMES:
The behavior measures of food texture related properties of commonly consumed foods | Through study completion, an average of 3hours visit per week
  The eating rate was measured and the bite size was quantified

CONTACTS AND LOCATIONS:
Overall Officials: Monica Mars, PhD, Study Chair — Wageningen University

REFERENCES:
- [Derived] van Langeveld AWB, Teo PS, Mars M, Feskens EJM, de Graaf C, de Vries JHM. Evaluation of dietary taste patterns as assessed by FFQ against 24-h recalls and biomarkers of exposure. Eur J Clin Nutr. 2019 Jan;73(1):132-140. doi: 10.1038/s41430-018-0300-1. Epub 2018 Sep 25. PMID 30254242